CLINICAL TRIAL: NCT01525667
Title: A Phase I/II, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Intramuscular Injections of Allogeneic PLX-PAD Cells for the Regeneration of Injured Gluteal Musculature After Total Hip Arthroplasty
Brief Title: Safety and Efficacy of IM Injections of PLX-PAD for the Regeneration of Injured Gluteal Musculature After Total Hip Arthroplasty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pluristem Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLX-PAD 1301-01
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-01

CONDITIONS: Total Hip Arthroplasty; Muscle Injury
Keywords: THA; Muscle injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 150M PLX-PAD (Experimental): Single course, multiple IM injections
  Interventions: Biological: 150M PLX-PAD
- 300M PLX-PAD (Experimental): Single course, multiple IM injections
  Interventions: Biological: 300M PLX-PAD
- Placebo (Placebo Comparator): Single course, multiple IM injections
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 150M PLX-PAD — Single course, multiple IM injections
  Arms: 150M PLX-PAD
Biological: 300M PLX-PAD — Single course, multiple IM injections
  Arms: 300M PLX-PAD
Biological: Placebo — Single course, multiple IM injections
  Arms: Placebo

SUMMARY:
Local administration of PLX-PAD single dose, intra-muscular injection for the regeneration of injured gluteal musculature after Total Hip Arthroplasty (THA).

DETAILED DESCRIPTION:
One of the main problems when performing THA via the standard transgluteal approach is the necessary injury of the gluteus medius muscle. The consecutive decrease of contractile muscle substance and the substitution by scar tissue leads to functional deficits of the pelvic-stabilizing musculature with an insufficiency limp in a large number of patients. In the long run the lack of musculature leads to a decrease in bone substance at the insertion sites of the gluteal muscles of the proximal femur. The present study has the aim of establishing a new therapy for iatrogenic gluteal muscle damage. The hypothesis of the present proposal is that intra-muscular (IM) injection of PLX-PAD into the iatrogenically injured gluteus medius muscle after THA results in an improved regeneration of the skeletal muscle tissue and consecutively in an improved functional outcome.

Subjects will be assigned to receive one of the two targeted doses of PLX-PAD or placebo. On the treatment day, after suturing the gluteus medius muscle PLX-PAD or placebo will be applied directly to the site of laceration.

Patients will be followed up for efficacy assessment up to week 26 and for safety assessment (Adverse events, vital signs, ECG, routinf lab and immunological testing) up to week 52 after THA. Patients will be phoned at week 104 in order to inquire about the occurence of new cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 50 to 75 years of age
2. Scheduled THA
3. ASA Score ≤ 3
4. Signed written informed consent

Exclusion Criteria:

1. Muscle diseases
2. Severe neurological diseases
3. Opioid long term medication
4. Pain chronification > stadium II of Gerbershagen
5. Immunosuppression due to illness or medication
6. Ankylosing spondylitis
7. History of ectopic bone formation of any localisation
8. Exclusion criteria for MRI (pace maker, defibrillator, ferromagnetic intracerebral clips)
9. Uncontrolled hypertension (defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 200 mmHg during screening)
10. Life-threatening ventricular arrhythmia or unstable angina - characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged
11. ST segment elevation myocardial infarction and/or TIA/CVA within three (3) months prior to enrollment. Subjects with severe congestive heart failure symptoms (i.e. NYHA Stage IV)
12. Subject has malignancy undergoing treatment including chemotherapy, radiotherapy or immunotherapy
13. Body Mass Index (BMI) of 35 Kg/m2 or greater
14. Known allergies to protein products (horse or bovine serum, or porcine trypsin) used in the cell production process
15. Known HIV, syphilis at time of screening
16. Known active Hepatitis B, or Hepatitis C infection at the time of screening
17. Pregnant or breast-feeding women or women of childbearing potential not protected by an effective contraceptive method of birth control (defined as pearl index < 1)
18. In the opinion of the investigator, the subject is unsuitable for cellular therapy
19. Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s)
20. Subjects who are legally detained in an official institute

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Perka, MD, Principal Investigator — Charité Universitätsmedizin Berlin, Dept. Of Orthopedic Surgery, Charitéplatz 1, 10117 Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- PLX-PAD Low Dose: 150M PLX-PAD : Single treatment, multiple injections
- PLX-PAD High Dose: 300M PLX-PAD : Single treatment, multiple injections
- Placebo: Placebo: Single treatment, multiple injections
Period: Overall Study
Arm/Group | PLX-PAD Low Dose | PLX-PAD High Dose | Placebo
Started | 7 | 6 | 7
Completed | 7 | 6 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PLX-PAD Low Dose: PLX-PAD low dose: Single treatment, multiple injections
- PLX-PAD High Dose: PLX-PAD high dose: Single treatment, multiple injections
- Total: Total of all reporting groups
Arm/Group | PLX-PAD Low Dose | PLX-PAD High Dose | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 9
  >=65 years | 4 | 4 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (5.9) | 64.5 (7.4) | 64.3 (6.4) | 64.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 6 | 10
  Male | 4 | 5 | 1 | 10
Region of Enrollment [Number; unit: participants]
  Germany | 7 | 6 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Day 0 to Week 26 in the Maximal Voluntary Isometric Contraction (MVIC) Moment of the Injured Side to Assess Gluteus Medius Strength.
Description: Change from Visit 2 (Day 0) to Week 26 in the maximal voluntary isometric contraction (MVIC) moment of the injured side as measured by isometric dynamometry to assess Gluteus Medius force strength.
Time Frame: Day 0 to Week 26
Measure: Least Squares Mean (Standard Error); unit: Newtons
Arm/Group | PLX-PAD Low Dose | PLX-PAD High Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 7
Newtons | 31.17 (6.97) | 20.36 (7.61) | 5.43 (6.46)
Statistical Analysis 1: Comparison: PLX-PAD Low Dose vs Placebo; Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis; Least Square Means (LSM) Difference = 25.74, 95% CI 2-sided [7.61 to 43.86], Standard Error of Mean 8.94 — LSM difference =LSM Low dose - LSM Placebo
Statistical Analysis 2: Comparison: PLX-PAD High Dose vs Placebo; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis; Least Square Means (LSM) difference = 14.93, 95% CI 2-sided [-7.12 to 36.99], Standard Error of Mean 10.80 — LSM difference= LSM High Dose - LSM Placebo

2. Secondary Outcome: Change From Day 0 to Week 26 in Muscle Volume.
Description: Change from Visit 2 (Day 0) to Week 26 in Muscle Volume as Measured by MRI.
Time Frame: Day 0 to Week 26
Measure: Least Squares Mean (Standard Error); unit: mm3
Groups:
- 150M PLX-PAD: PLX-PAD low dose: Single treatment, multiple injections
- 300M PLX-PAD: PLX-PAD high dose: Single treatment, multiple injections
Arm/Group | 150M PLX-PAD | 300M PLX-PAD | Placebo
Number analyzed (Participants) | 7 | 6 | 7
mm3 | 24.42 (4.18) | 15.62 (4.91) | 6.39 (4.35)
Statistical Analysis 1: Comparison: 150M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LSM Difference = 18.03, 95% CI 2-sided [6.03 to 30.02], Standard Error of Mean 5.97
Statistical Analysis 2: Comparison: 300M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis; LSM difference = 9.23, 95% CI 2-sided [-4.72 to 23.17], Standard Error of Mean 6.91

3. Secondary Outcome: Change From Day 1 to Week 12 in Mean Fiber Diameter.
Description: Change from Visit 3 (Day 1) to Week 12 in Mean Fiber Diameter as Measured by Muscle Biopsy.
Time Frame: Day 1 to Week 12
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | 150M PLX-PAD | 300M PLX-PAD | Placebo
Number analyzed (Participants) | 7 | 6 | 7
microns | 1.25 (3.27) | 0.28 (3.23) | -5.21 (3.24)
Statistical Analysis 1: Comparison: 150M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.19, ANCOVA; LSM Difference = 6.45, 95% CI 2-sided [-3.50 to 16.41], Standard Error of Mean 4.64
Statistical Analysis 2: Comparison: 300M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.25, ANCOVA; LSM difference = 5.49, 95% CI 2-sided [-4.29 to 15.26], Standard Error of Mean 4.56

4. Secondary Outcome: Change From Day 0 to Week 26 in the Ratio of Injured to Contralateral Pelvic Shift .
Description: Change from Visit 2 (Day 0) to Week 26 in the Ratio of Injured to Contralateral Pelvic Shift as Measured by Gait Analysis
Time Frame: Day 0 to Week 26
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 150M PLX-PAD | 300M PLX-PAD | Placebo
Number analyzed (Participants) | 7 | 6 | 7
Ratio | 0.43 (0.13) | 0.28 (0.14) | 0.27 (0.13)
Statistical Analysis 1: Comparison: 150M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.4, Mixed Models Analysis; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.21 to 0.53], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: 300M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.96, Mixed Models Analysis; Mean Difference (Net) = 0.011, Standard Error of Mean 0.20

5. Secondary Outcome: Change From Day 0 to Week 26 in the Visual Analog Scale (VAS) Pain Score.
Description: Visual Analog Scale (VAS) Pain Score ranges from 0 mm (no pain) to 100 mm (worse possible pain)
Time Frame: Day 0 to Week 26
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 150M PLX-PAD | 300M PLX-PAD | Placebo
Number analyzed (Participants) | 7 | 6 | 7
mm | -31.76 (5.90) | -37.87 (6.53) | -48.57 (5.97)
Statistical Analysis 1: Comparison: 150M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; LSM difference = 16.81, 95% CI 2-sided [0.16 to 33.47], Standard Error of Mean 8.37
Statistical Analysis 2: Comparison: 300M PLX-PAD vs Placebo; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis; LSM difference = 10.70, 95% CI 2-sided [-7.26 to 28.65], Standard Error of Mean 9.01

ADVERSE EVENTS:
Time Frame: Data were collected for total period of 1 year.
Arm/Group | 150M PLX-PAD | 300M PLX-PAD | Placebo
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150M PLX-PAD (N=7) | 300M PLX-PAD (N=6) | Placebo (N=7)
HUMERAL HEAD FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
PERIURETHRAL CYST (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150M PLX-PAD (N=7) | 300M PLX-PAD (N=6) | Placebo (N=7)
Breath odour (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (7) | 3 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Post procedural swelling (Injury, poisoning and procedural complications) | 3 (3) | 3 (4) | 2 (4)
Suture related complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No